CLINICAL TRIAL: NCT03964623
Title: Impact of Nicotine on Retinal Vascularization (Tabaret)
Brief Title: Impact of Nicotine on Retinal Vascularization
Acronym: TABARET
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: VVR_2019_5
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Tabagism
Keywords: OCT-A; smokers; vapers; non-smokers/non-vapers; nicotine; retinal micro-vascularization
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- smokers
  Interventions: Diagnostic Test: OCT-A (Optical Coherence Tomography)
- vapers
  Interventions: Diagnostic Test: OCT-A (Optical Coherence Tomography)
- non smokers/non vapers
  Interventions: Diagnostic Test: OCT-A (Optical Coherence Tomography)

INTERVENTIONS:
Diagnostic Test: OCT-A (Optical Coherence Tomography) — Included patients will have an OCT-A and will be questioned about their nicotine intake, their background and taking an oral conception

SUMMARY:
The main hypothesis is the nicotine is associated with a modification of retinal micro-vascularization.

Patients will be recruited during their ophthalmologic consultation at the Rothschild Foundation, an OCT-A will be realized and data relating to medical history, oral contraceptive intake and nicotine consumption via cigarette or e-cigarette data will be collected.

The objective is to seek an association between retinal vascular density and inhaled nicotine intake.

ELIGIBILITY:
Inclusion criteria

* For group of smokers: Patient reporting active smoking for at least 3 months and at least 1 cigarette per day on average over a week
* For group of vapers : Patient using exclusively the electronic cigarette with a nicotine level of more than 6mg/ml for at least 3 months and at least 1 times per day on average over a week.
* For group of no-smokers no-vapersNon-smoking and no vaping, for more than 6 months

Non-inclusion criteria:

* Caffeine intake within 2 hours prior to the OCT-A exam
* ametropia greater than + 3 dioptres of hyperopia or-3 dioptres of myopia
* astigmatism greater than 2 dioptres
* Known retinal or retina vascular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People presenting to an ophthalmologic consultation at the Foundation Rothschild will be included in one of the 3 groups: smokers, non-smokers/non-vapers or vapers if they meet the inclusion and non-inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Density of retinal vascular Plexus (quantitative variable expressed as a percentage) using OCT-A. | At the inclusion consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No